CLINICAL TRIAL: NCT06195969
Title: Automated Instant Message-guided Hypertension Management Intervention Among Stroke Survivors: a Pilot Trial
Brief Title: Instant Message-guided Hypertension Management Intervention Among Stroke Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HTN2023
Record Dates: First submitted 2023-12-08; First posted 2024-01-08 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Stroke; Hypertension; Lifestyle Modifications
Keywords: Stroke; Hypertension Management
MeSH Terms: conditions — Stroke; Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants in intervention group will receive the EMI for 4 weeks. Based on the steps of mobile message development recommended by Abroms, et al. , we will develop a message content library and protocol for EMI delivery.
  Interventions: Behavioral: automated instant message-guided hypertension management intervention group
- Control group (No Intervention): The control group will receive instant messages about general stroke management including hypertension management from the Hospital Authority of HK SAR Government website, which is open to the public (https://www21.ha.org.hk/smartpatient/SPW/en-US/Disease-Information/Disease/?guid=29ac1219-3d68-4378-a2bd-09e111da3650), with reminder text messages of importance follow-up surveys.

INTERVENTIONS:
Behavioral: automated instant message-guided hypertension management intervention group — Participants in intervention group will receive the EMI for 4 weeks. Based on the steps of mobile message development recommended by Abroms, et al., we will develop a message content library and protocol for EMI delivery
  Arms: Intervention group

SUMMARY:
This pilot and feasibility study aims to develop an automated instant message-delivered intervention (i.e., EMI) for hypertension management in stroke survivors, and to investigate the feasibility and effectiveness of the intervention.

DETAILED DESCRIPTION:
Intervention group:

Participants in intervention group will receive the EMI for 4 weeks. Based on the steps of mobile message development recommended by Abroms, et al., we will develop a message content library and protocol for EMI delivery.

1. Message contents: The message content library will consist of two parts: 1. brief stroke and hypertension education messages (mandatory), and 2. lifestyle modification messages (optional).
2. Message delivery

   * Regular messages: The messages in the two parts will be sent regularly to each participant. As personalisation is a core process subject to behavioural changes, the content, frequency, and timing of the messages will be determined based on participants' preferences. To save labour and increase efficiency, we will develop a message 'scheduler' program. We will pre-set the message scheduler, which will then automatically send out content to participants according to their preferences. The development of the program is highly useful particularly in cases which participants prefer to receive messages during non-office hours.
   * Nurse-led real-time support messages (chat-type): Chat-based nurse support will be given to the participants as an extension of the regular messages. However, the participants will be informed beforehand that the nurse will only play a supportive role and will not provide formal care. The number of the chat messages will not be limited, but the nurse-led real-time support messages will only be provided during working hours (i.e., 9am-6pm) on weekdays to limit the nurse RA's workload.

Control Group:

The control group will receive one instant message about general stroke management including hypertension management from the Hospital Authority of HK SAR Government website (https://www21.ha.org.hk/smartpatient/SPW/en-US/Disease-Information/Disease/?guid=29ac1219-3d68-4378-a2bd-09e111da3650), which is open to the public.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stroke (ICD-10 codes: I60-I69)
* Diagnosis of hypertension and antihypertension medication
* Aged ≥18
* Able to read and communicate in Chinese (Cantonese or Putonghua)
* Able to use text messaging function on mobile phones
* MoCA 5-minute Protocol (cognitive screen) ≥14 (Equivalence to MMSE ≥ 21)

Exclusion Criteria:

* Currently receiving active stroke care in acute or post-acute inpatient settings
* Has diagnosis of psychiatric disease or is currently taking psychotropic drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-11-13 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-01-12 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure | 4 weeks
  A validated blood pressure monitor will be used to evaluate the participants' blood pressure. A higher systolic blood pressure number indicates higher blood pressure.
Diastolic blood pressure Diastolic blood pressure | 4 weeks
  A validated blood pressure monitor will be used to evaluate the participants' blood pressure. A higher diastolic blood pressure number indicates higher blood pressure.

SECONDARY OUTCOMES:
Self-efficacy (Stroke Self-Efficacy Questionnaire) | 4 weeks
  Each item was scored on an 11-point scale (0 "not at all confident" to 10 "very confident"). The total score is calculated by summing up the score of all items (range 0-130). High scores indicate greater self-efficacy.
Quality of life (EuroQol 5-dimension 5-level questionnaire) | 4 weeks
  The EQ-5D-5L is a self-assessed, health related, quality of life questionnaire. The scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Higher scores indicate worse quality of life.
Feedback on Instant Message-Guided Hypertension Management Intervention | 4 weeks
  We will conduct a broad assessment of participant feedback in this blood pressure management program, covering aspects such as the perceived value of the program. Each area will be evaluated using a 5-point Likert scale, where higher scores will consistently indicate more positive assessments across all metrics.
Self-care of high blood pressure (SC-HI) | 4 weeks
  The SC-HI is a 23-item measure of self-care maintenance, monitoring, and management appropriate for persons with chronic HTN. Each dimension is scored on a scale ranging from 0 to 100, with higher scores reflecting more effective self-care behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Jung Jae Lee, Principal Investigator — School of nursing, the University of Hong Kong
Locations (7):
- Hong Kong (7):
  - Hong Kong PHAB Association, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - Shatin Hospital, Hong Kong
  - Southern District Elderly Community Centre, Hong Kong
  - The Hong Kong Society for Rehabilitation, Hong Kong
  - Tung Wah Hospital, Hong Kong
  - United Christian Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: No